CLINICAL TRIAL: NCT02982239
Title: Recovery Enhancement and Sleep Training (REST): Sleep and Mental Well-Being in Student Athletes
Brief Title: Recovery Enhancement and Sleep Training
Acronym: REST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Collegiate Athletic Association - NCAA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1605615210
Record Dates: First submitted 2016-10-25; First posted 2016-12-05 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2016-11

CONDITIONS: Sleep; Performance; Mental Health; Stress; Anxiety
MeSH Terms: conditions — Psychological Well-Being; Anxiety Disorders | interventions — Fitness Trackers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Intervention (Other): N=20 Participants received fitness tracker, information session, a link to complete a daily sleep diary, intermittent text messages that included adherence reminders, encouraging statements, and tips for improving sleep. Daily monitoring with sleep diaries, daily monitoring of sleep tracker sync activity and regret lottery for 10 weeks
  Interventions: Behavioral: Sleep Diary; Device: Fitness tracker; Other: Information Session; Behavioral: Text messages
- Sleep Intervention plus Tech (Other): N=20 Participants received fitness tracker, LED light, Blue-blocking glasses along with information session, a link to complete a daily sleep diary, intermittent text messages that included adherence reminders, encouraging statements, and tips for improving sleep. Daily monitoring with sleep diaries, daily monitoring of sleep tracker sync activity and regret lottery for 10 weeks.
  Interventions: Behavioral: Sleep Diary; Device: Fitness tracker; Device: Blue-Blocking Glasses; Device: LED light; Other: Information Session; Behavioral: Text messages

INTERVENTIONS:
Behavioral: Sleep Diary — All 40 chosen students will be provided a link to complete a daily sleep diary for 10 weeks. Sleep diary will assess activity before bed, bedtime, time to fall asleep, number of awakenings, time awake after sleep onset, time out of bed, time of final awakening, perceived sleep quality. Diary also asks about naps taken during the day, caffeine and tobacco consumption, and an additional space for open-ended comments from the participant.
Device: Fitness tracker — All 40 chosen students will receive a fitness tracker. The fit bit will estimate sleep and physical activity as well as adherence to the program. participants will have access to their own data. Data will also be monitored from the lab using Fitabase which provides access to day, hour, and minute-level resolution of data for steps taken, intensity class, calories burned, and sleep (length, movement, and quality).
Device: Blue-Blocking Glasses — Half of the 40 chosen students (N=20) will be provided with blue blocking glasses. The blue-blocking glasses will ensure that blue light from electronic devices will not interfere with circadian rhythm or sleep onset, and allow students to fall asleep earlier.
  Arms: Sleep Intervention plus Tech
Device: LED light — Half of the 40 chosen students (N=20) will be provided with a bright LED light. The bright LED light will provide bright blue light in the morning to help students wake and an amber light to promote earlier bedtimes.
  Arms: Sleep Intervention plus Tech
Other: Information Session — all 40 participants will attend a 1-hour information session about sleep delivered by the PIs, to be followed by a 1-hour Q&A period.
  Peer educators will receive and extra 1-hour training session on how to handle questions and when to refer back to the PIs.
  Other Names: Educational session
Behavioral: Text messages — All participants will receive text messages in the evening that will include adherence reminders, encouraging statements, and tips for improving sleep. Messages will be randomized, with no more than 3 messages of any type per week. Messages will serve as a cue to action without being overly repetitive or predictable.

SUMMARY:
Evidence suggests that student athletes frequently experience sleep problems and are aware of the impact of sleep loss on mental and physical outcomes. As such, student athletes are motivated to improve sleep quality in order to improve their outcomes for overall athletic performance. This study will consist of two parts. The first part will be a survey. Fall athletes arrive in the summer, and Part 1 will invite 200 of these athletes to complete a survey within the first week of their arrival on campus. The survey will assess multiple domains of student-athlete health, namely, sleep duration and quality, mood and depression, stress, and mental and physical well-being. The responses to the survey will be confidential, and students will be compensated for the survey. At the end of the semester, students will be invited to complete the survey again.

Part 2 is an intervention. 40 of the 200 students will be chosen to participate in the intervention, based on predetermined criteria. The intervention will include an information session where students may ask questions. Students will be sent text message reminders about adherence to the program and will be asked to monitor their sleep quality with sleep diaries. The intervention will consist of the half of the 40 chosen students, (20 students), who will be provided with blue blocking glasses, a bright light-emitting diode (LED) light, and a fit bit. Please note that all of these items are commercially available and are not meant to be used to treat or prevent human illness nor injury and do not require FDA oversight. The blue-blocking glasses will ensure that blue light from electronic devices will not interfere with circadian rhythm or sleep onset, and allow students to fall asleep earlier. The bright LED light will provide bright blue light in the morning to help students wake and an amber light to promote earlier bedtimes. The Fitbit will estimate sleep and physical activity as well as adherence to the program.

DETAILED DESCRIPTION:
Student athletes face many challenges to their ability to maintain healthy mental and physical well-being. The college experience is associated with a number of physiologic, social, and environmental stressors that can exert long-term effects on an individual's future health and quality of life. In addition, unique demands of student-athletes, including academic, physical performance, scheduling, and travel demands, all represent additional stressors that interact to produce in poorer outcomes.

Insufficient sleep duration and poor sleep quality have been increasingly identified as important risk factors for physical and mental well-being, especially among young adults. For example, insufficient and/or poor quality sleep is strongly associated with the development of cardiometabolic disease risk factors, obesity, depression, anxiety disorders, alcohol use, other substance use, poorer academic performance, and reduced mental well-being, in addition to poorer athletic performance.

Data from a recent PAC12 conference report shows that 2/3 of students indicated that lack of flexible time is the hardest thing about being an athlete, more than academic work. Further, students identified sleep as the first thing that their athletic time commitments kept them from doing, 77% felt that they got less sleep than non-athletes, and >50% indicated that they would use an extra hour to catch up on sleep. In 2015 data from the American College Health Association, (1) 29% of student athletes report significant sleep difficulties, (2) 40% reported getting enough sleep on only ≤3 nights, (3) 10% reported no problems with daytime sleepiness, (4) >15% reported sleepiness to be at least "a big problem," (5) >25% reported extreme difficulty falling asleep ≥3 nights/week (consistent with a diagnosis of insomnia), and (6) >50% reported that sleep problems impacted academic performance. Thus, student-athletes frequently experience sleep problems, they recognize the impact of sleep loss, and they are likely motivated to improve sleep. These data are consistent with data from professional athletes, whose overall sleep quality is poorer than non-athletes.

Taken together, sleep is an aspect of health that is implicated in many of the most salient mental and physical outcomes among college athletes. Despite this, obtaining sufficient sleep represents one of the greatest challenges facing student athletes. No programmatic approaches have been able to address this problem.

Accordingly, the proposed study aims to develop and assess the benefits of a novel sleep health intervention targeted at student-athletes. This intervention will be assessed with and without the assistance of tools to aid in tracking sleep and adjusting to difficult schedules in order to evaluate the utility of those approaches.

The purpose of this research study is to develop and assess the benefits of a novel sleep health intervention targeted at student-athletes.

Overall objectives AIM 1: Assess cross-sectional relationships among sleep, circadian preference, and outcomes including overall mental health, stress, mood, anxiety, social functioning, and physical well-being.

AIM 2: Determine whether a simple sleep health intervention, with and without the aid of technology, is associated with improvements in mental and physical well-being.

Primary outcome variable(s) AIM 1: depression score, stress score, mental well-being score, anxiety score, and physical well-being score AIM 2: changes in AIM 1 outcomes Secondary outcome variable(s) Academic stress, physical performance, substance use, health behaviors, soft tissue injuries, missed practices, academic performance

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate
* Participation as a student-athlete during the entirety of their season
* No medical conditions that would preclude them from participating (assessed by self-report)
* Age ≥18 years

Exclusion Criteria:

* Freshmen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2017-01-05 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Student-athletes were recruited over the summer and through the first 2 weeks of the 2015 Fall semester, as they arrived on campus. Recruitment was accomplished through flyers, referrals from athletics staff, and in-person recruitment among athletes at on campus athletic facilities.
Pre-assignment Details: All students who completed the survey were eligible for the intervention study, though selection was targeted to those with sleep complaints.
Groups:
- Intervention- No Tech: Participants received fitness tracker, information session, a link to complete a daily sleep diary, intermittent text messages that included adherence reminders, encouraging statements, and tips for improving sleep. Daily monitoring with sleep diaries, daily monitoring of sleep tracker sync activity and regret lottery for 10 weeks
- Intervention -Tech: Participants received fitness tracker, LED light, Blue-blocking glasses along with information session, a link to complete a daily sleep diary, intermittent text messages that included adherence reminders, encouraging statements, and tips for improving sleep. Daily monitoring with sleep diaries, daily monitoring of sleep tracker sync activity and regret lottery for 10 weeks.
Period: Overall Study
Arm/Group | Intervention- No Tech | Intervention -Tech
Started | 20 | 20
Completed | 17 | 18
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Participants received fitness tracker, information session, a link to complete a daily sleep diary, intermittent text messages that included adherence reminders, encouraging statements, and tips for improving sleep. Daily monitoring with sleep diaries, daily monitoring of sleep tracker sync activity and regret lottery for 10 weeks
- Total: Total of all reporting groups
Arm/Group | Intervention | Intervention -Tech | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.56 (0.97) | 20.55 (0.93) | 20.55 (0.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Pittsburgh Sleep Quality Index ( PSQI)
Description: Change in Pittsburgh Sleep Quality Index (PSQI) score at the end of the 10-week intervention. The PSQI global score has a possible range of 0-21 points. A total score of 5 or above indicates overall poor sleep quality.
Time Frame: Change from baseline to post-intervention, around 10 weeks after baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Intervention -Tech
Number analyzed (Participants) | 17 | 18
units on a scale
  Baseline | 4.941176471 (2.9041046) | 6.555555556 (3.329409455)
  Post-intervention | 4.647058824 (2.84914848) | 5.833333333 (2.7917947)

2. Primary Outcome: Insomnia Severity Index (ISI)
Description: Change Insomnia Severity Index (ISI) score at the end of 10-week intervention. The Insomnia Severity Index is a frequently-used questionnaire to measure insomnia symptoms. Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
Time Frame: Change from baseline to post intervention, around 10 weeks after baseline
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention- No Tech | Intervention -Tech
Number analyzed (Participants) | 17 | 18
scores on a scale
  Baseline | 5.529411765 (4.862068066) | 7.5 (3.944467458)
  Post-intervention | 5.176470588 (4.034775305) | 5.266666667 (3.954503159)

3. Primary Outcome: Centers for Disease Control (CDC)l and Prevention Health-Related Quality of Life Scale (HRQOL)
Description: Change in CDC Health-Related Quality of Life Scale (HRQOL) score at the end of 10-week intervention. Health-related quality of life (HRQOL) is an individual's or a group's perceived physical and mental health over time. Unhealthy days are an estimate of the overall number of days during the previous 30 days when the respondent felt that either his or her physical or mental health was not good. Healthy days are the positive complementary form of unhealthy days. Healthy days estimates the number of recent days when a person's physical and mental health was good (or better) and is calculated by subtracting the number of unhealthy days from 30 days.
Time Frame: Change from baseline to post intervention, around 10 weeks after baseline
Measure: Mean (Standard Deviation); unit: Days out of 30
Arm/Group | Intervention | Intervention -Tech
Number analyzed (Participants) | 17 | 18
Days out of 30
  unhealthy mental health days Baseline | 6.176470588 (10.30919065) | 7.555555556 (8.958874813)
  unhealthy Physical health days Baseline | 5.411764706 (9.695738906) | 3.944444444 (6.803737919)
  unhealthy mental health days Post-Intervention | 6.411764706 (8.000459546) | 4.611111111 (5.699730529)
  unhealthy physical health days Post-Intervention | 6.352941176 (9.512762325) | 6.833333333 (9.173170598)

4. Primary Outcome: Centers for Epidemiological Studies Depression Scale (CESD)
Description: Change in Centers for Epidemiological Studies Depression Scale (CESD) score at the end of 10-week intervention. Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.
Time Frame: Change from baseline to post intervention, around 10 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Intervention -Tech
Number analyzed (Participants) | 17 | 18
score on a scale
  CESD total score Baseline | 8.294117647 (6.45914764) | 10.16666667 (7.957608272)
  CESD total score Post-Intervention | 9.470588235 (8.147987843) | 7.333333333 (6.962082177)

5. Primary Outcome: Perceived Stress Scale (PSS)
Description: Change in Perceived Stress Scale (PSS) score at the end of the 10-week intervention.The PSS is comprised of 14 items intended to measure how unpredictable, uncontrollable, and overloaded individuals find their life circumstances.Participants rate items on a 5-point Likert scale, ranging from 0 - "Never" to 4 - "Very often." Scores range from 0-56 higher scores indicate greater perceived stress.
Time Frame: Change from baseline to post intervention, around 10 weeks after baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention- No Tech | Intervention -Tech
Number analyzed (Participants) | 17 | 18
score on a scale
  Baseline | 21.52941176 (7.072107598) | 21.27777778 (5.706606652)
  Post-intervention | 23.05882353 (7.386394488) | 19.11111111 (7.379533613)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Intervention | Intervention -Tech
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Since this is considered a pilot study and is likely underpowered, the primary outcomes were assessed for change over time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No